CLINICAL TRIAL: NCT02255981
Title: ¿Es Util la Acupuntura en la Degeneracion Macular? Prospective Study of Efficacy of Acupuncture in Macular Diseases
Brief Title: Efficacy of Acupuncture in Macular Diseases
Acronym: AMAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escuela Neijing (Other)
Responsible Party: Principal Investigator, Dra. Luz Helena Gutiérrez C, Luz Gutierrez Physician, MPH, Escuela Neijing, Research Coordinator., Escuela Neijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neijing Ophthalmology
Record Dates: First submitted 2014-09-25; First posted 2014-10-03 (Estimated); Results first posted 2020-04-01 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Age-related Macular Degeneration; Stargardt Disease; Macular Dystrophy
Keywords: macular degeneration, acupuncture, OCT, Stargardt, dystrophy
MeSH Terms: conditions — Macular Degeneration; Stargardt Disease; Ornithine Carbamoyltransferase Deficiency Disease | interventions — Acupuncture Therapy; Massage; Medicine, Chinese Traditional

STUDY DESIGN:
Intervention Model Description: Interventional, no randomized, no masking
Masking Description: Masking is neither accurate nor reliable in a procedure such as acupuncture or massage.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acupuncture group (Experimental): Acupuncture and massage Therapy of Traditional Chinese Medicine (acupuncture and Massage) for 24 months
  .
  Interventions: Other: Acupuncture and massage

INTERVENTIONS:
Other: Acupuncture and massage — Treatment consists in to put needles on specific points of skin one day each week initially, then with longer spaces of time according to improvement.A total of 11 Chinese needles stainless steel, 25 x 40 were used by manual insertion and left for 12-15 minutes.
  Periocular massage is taught and is practiced daily by the patient him or herself.
  Other Names: Traditional Chinese Medicine:( TCM); acupuncture chinese style

SUMMARY:
This is a single-arm study designed to assess the efficacy of acupuncture (Traditional Chinese Medicine) for chronic macular diseases of several types. All participants received acupuncture and massage and there is not a placebo group because it is not considered a good form to evaluate in Chinese Medicine due to, acupuncturing being a procedure is not as blind as is desired. As a control of the results in this trial, the outcomes could be contrasted against those reported in known medical publications and against expectations of the progress of the damage without treatment.

DETAILED DESCRIPTION:
Background.

WHO has included retinal diseases between conditions treatable by acupuncture and Traditional Chinese Medicine (TCM) has been used for retinal diseases in hospitals of China and in other parts of the world many years ago. Acupuncture and periocular massage act stimulating the vital energy to restore the normal function of the body.

Currently, most common treatments in Western Medicine, anti-VEGF, only are indicated for less than 10 percent of cases, which are the wet form or neovascular of AMD (NV-AMD) and they have restrictions for use, additionally, their cost and requirements are limiting for populations in all countries.

Objectives. The primary purpose of this study is to confirm the objective response among subjects with macular diseases treated with acupuncture and massage. The results of conventional treatment are published in similar trials and some of our patients have had intraocular injections previously.

It is important to feature the affordability of this therapy for low-income populations that do not have specialists or facilities nearby or for many governments that complain about the huge burden of the treatment of there diseases. In Colombia, the average cost of each intraocular injection by the time of this trial was about US 3.500 and it can be repeated every month, it requires a retina specialist and a surgical room, that is out of reach for many people in the country.

We did not calculate the costs of our treatment because the research team did voluntary labor, and the devices are at a very low cost, about US 0.50 in each session. Acupuncture treatment does not require special facilities as surgical rooms required in treatments with intraocular injections. The participants were not paid, they came from different economic conditions, some better, others from poorest neighborhoods or some from the rural areas.

This study includes 3 phases: Selection, Treatment, and Follow-up phases.

The selection phase included confirmed diagnosis by clinical register and OCT, Ophthalmologic assessment, and consent of the patient.

Macular diseases. In this trial, some patients had NV AMD in one or both eyes, dry AMD, myopic maculopathy or Stargardt disease. For TCM it is possible to treat all as damage of similar category.

Why no control group. There was no control group due to ethical reasons, leave the impairment without treatment in these mostly very sad persons. The second reason is the well-known difficulty to mask a procedure like acupuncture. another third reason is the possibility to contrast the results of this trial with those of similar studies conducted in eyes with conventional treatment.

In the phase of treatment, Patients received a session of acupuncture according to a standard protocol of points, and a periocular massage that was taught to the patient to be self-performed daily. The acupuncture sessions were scheduled every week initially, the evaluation of response was realized every 2 months by ophthalmologic exam and was asked to participants an optical coherence tomography (OCT) that would be realized every 6 months. Depending on the results of ophthalmologic assessment the sessions were extended gradually to every 2, 3, 5 until 13 weeks. Although tomographic assessments had been scheduled every 6 months, only a few of the participants accomplish with that due to economic limitations. Treatment continued until 24 months

All patients in the follow-up phase of this trial were monitored according to the Safety Follow-up protocol and the defined procedures and evaluations.

The final results were collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* • Clinical diagnosis of Macular Disease.

  * The patient must accept treatment with acupuncture

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-03; Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luz H Gutierrez, MD, MPH, Principal Investigator — Escuela Neijing Colombia; Jose L Padilla, MD, Study Director — Hispano American Acupuncture Association-Beijing 84, Madrid, Spain; José R Gutiérrez, MD, Opht, Study Chair — Sociedad Colombiana de Oftalmología; Libia V Ferrer, Tech TCM, Study Chair — Escuela Neijing Colombia; Sergio L Pineda, Study Chair — Escuela Neijing Colombia
Locations (2):
- Colombia (2):
  - IPS Fundación Neijing, Guarne, Antioquia
  - IPS Fundación Neijing, Medellín, Antioquia

IPD SHARING:
Plan to Share IPD: Yes
sex, age, ophthalmologic diagnostic data (medical examination, images) diagnostic signs on Traditional Chinese Medicine (TCM), number of sessions, visual outcome, hazards, previous treatment. Individual participant data that underlie the results reported will be shared after deidentification
Supporting Information: CSR
Time Frame: Inmediate following publication and no end term.
Access Criteria: Any

REFERENCES:
- [Result] Gutierrez L, Pineda S, Gutierrez R, Ferrer L. Acupuncture in Macular Diseases (AMAD) No published yet

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Project was announced to ophthalmologists asking them to refer patients. Very few arrived by reference and most entered by personal interest. Study was conducted in Medical consultation site of Neijing School, in Medellín, Colombia The recruitment period was between April 2013 and May 2014.
Pre-assignment Details: 35 patients were eligible, 2 refused to participate, 29 completed follow up. There was not an assignment, all received the same treatment although the diagnostics comprised different forms of macular damage it was pre-specified to analyze them as a single group for the Outcomes 2 eyes were excluded: 1 blind and 1 with retinal detachment.
Units Other Than Participants: eyes
Groups:
- Acupuncture & Macular Damage: Intervention: Acupuncture (Traditional Chinese Medicine) and Massage: A total of 11 Chinese needles 25 x 40 were used by manual insertion. Periocular massage is teached and is practiced daily by the patient him or herself
  .
  Acupuncture Traditional Chinese Medicine (TCM): Treatment consist in to put needles on specific points of skin one day each week initially, then with longer spaces of time according to improvement.
Period: Overall Study
Arm/Group | Acupuncture & Macular Damage
Started | 33; 64 eyes (Both eyes of each patient were included except 2 that not were treatable)
Completed | 29; 56 eyes (2 eyes of the final 29 subjects were excluded.)
Not Completed | 4; 8 eyes
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: 35 patients met inclusion criteria, 33 consented to participate, 4 dropped off, 29 ended the 24 month period of treatment and observation
Arm/Group | Acupuncture & Macular Damage
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Change on Visual Acuity (VA) of the Treated Eyes From Baseline to the End of the Study
Description: The primary objective is to assess if acupuncture treatment is linked to a change in visual acuity (VA).
  VA was obtained by an ophthalmologic assessment at baseline and every two months until month 24. VA measurements were taken with the patient in a sitting position using a Snellen chart at a testing distance of 6 meters. The scale in Snellen is given in fractional numbers corresponding 20/20 to a normal vision at 20 ft or 6 meters. According to the World Health Organization, the normal vision is to 20/25, severe impairment corresponds to VA worse than 20/200 or legal blindness. Each fraction corresponds to a determined line of the chart in which all letters are correctly identified and the variation or gain is appreciated by the lines gained or lost by each eye.
  Improvement means a fraction better than initial, stable is no change in VA and lost is the VA worst than those of baseline.
Time Frame: Baseline, 2 months and every 2 months until month 24.
Population: The primary analysis includes only patients who completed the 24-month exam. The improvement in this outcome is measured on eyes which had a vision gain in lines of the Snellen chart.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Groups:
- Change in VA From Baseline to the End of Study: There were 13 patients with neovascular AMD in one or in both eyes. The total of eyes in this condition was 22 and the other 13 participants, had the dry form of AMD in one or both of his eyes, for a total of 23 eyes. This is not the sum of participants in each form of the disease because some of them had mixed conditions. Other 4 patients, 8 eyes, had macular dystrophy and 2 participants (3 eyes) had myopic degeneration. As the objective was not the comparison between them, it was prespecified analyze them together
Arm/Group | Change in VA From Baseline to the End of Study
Number analyzed (Participants) | 29
Number analyzed (Eyes) | 56
Eyes
  Eyes which improved VA | 36
  Eyes with stable VA | 16
  Eyes which lost VA | 4

2. Primary Outcome: Eyes With Change From Baseline to the End of the Study in Distance Vision According to Categories CIE 10 Based on Lines Seen on the Snellen Chart.
Description: Change in Visual Acuity was Measured by the Numbers of Lines seen on the Snellen Chart from baseline to the end of the trial. The measure was obtained by an ophthalmologic assessment on both eyes at the beginning of the study and every two months until month 24 using the best correction. VA measurements (lines in which all letters are correctly identified) were performed with the patient in a sitting position using a Snellen chart at a testing distance of 6 meters and the variation is appreciated by the lines gained or lost by each eye. The measure in Snellen is given in fractional numbers. Each fraction corresponds to a determined line of the chart corresponding VA 20/20 or 6/6 to a normal vision at 20 ft or 6 meters. The range of normal vision according to the WHO is to 20/25 ft or 6/10m, Mild means VA worse than 6/12, Moderate means VA worse than 6/18, Severe means VA worse than 6/60 that is "legal blindness". Blindness is considered VA worse than 3/60.
Time Frame: 24 months from baseline.
Population: All participants received the same treatment in a treat and extend regimen with an ophthalmological review every 2 months for 2 years. Data of VA from baseline to the end of the study were compared to assess Improvement or worsening. Improved means eyes with a better score of lines, stable means equal VA and worse is a loss of lines seen.
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Groups:
- VA Measured at Snellen Chart at the Beginning of the Study: In all participants, VA was measured at baseline. The category of visual impairment according to WHO, ICD-10 is presented below.
- VA Measured at Snellen Chart at the End of the Study: VA was measured by an ophthalmologist every 2 months. The numbers below are the final VA at 24 months from the beginning.
Arm/Group | VA Measured at Snellen Chart at the Beginning of the Study | VA Measured at Snellen Chart at the End of the Study
Number analyzed (Participants) | 29 | 29
Number analyzed (Eyes) | 56 | 56
Eyes
  Normal | 20 | 29
  Mild | 3 | 4
  Moderate | 9 | 8
  Severe | 19 | 10
  Blindness | 5 | 5

3. Primary Outcome: Change From Baseline in the Number of Letters Seen on the Early Treatment Diabetic Retinopathy Study (ETDRS) Eye Chart
Description: The ETDRS scale of letters is commonly used to report outcomes in AMD, for this reason, this score was chosen to compare outcomes with similar studies. Accepted tables for conversion from Snellen to ETDRS were used. 85 letters are equivalent to 20/20 and 0 letters correspond to 20/200. It can be meaningful to analyze the results in this trial in the context of similar trials using anti-VEGF, or reporting a visual loss in those cases that are not treatable.
Time Frame: Baseline and at end of study (up to 2 years)
Population: In AMD patients, some had a form in one eye and other in the fellow. "Improved" means the eyes which improved based on the number of letters gained in the ETDRS chart over the baseline and maintained for the end of the study. "Stable" if the number of letters is almost the same and "lost" if it was reduced.
Measure: Mean (Standard Deviation); unit: Letters on ETDRS scale
Units Other Than Participants: eyes
Groups:
- All Eyes Which Received Acupunture for 24 Months: The ETDRS scale of letters is commonly used to report outcomes in AMD, for this reason, this score was chosen to compare outcomes with similar studies. Accepted tables for conversion from Snellen to ETDRS were used.
  There were 22 eyes diagnosed with NV AMD, 23 eyes with no NV AMD, 8 eyes with macular dystrophy, and 3 eyes with Myopic degeneration. 2 eyes of all participants were excluded due to its status, one blind and one with retinal detachment. Although the observation collected the data for each macular disease form, the objective of the trial was not to compare between types of the disease and the results are grouped for the total of eyes.
Arm/Group | All Eyes Which Received Acupunture for 24 Months
Number analyzed (Participants) | 29
Number analyzed (eyes) | 56
Letters on ETDRS scale
  Letters seen at baseline | 41.5178 (33.7127)
  Letters seen at the end of study | 53.5714 (30.2450)
  Change from baseline | 14.3571 (18.8684)
Statistical Analysis 1: Comparison: All Eyes Which Received Acupunture for 24 Months; Besides that it is of interest to compare with the published studies outcomes, realized with anti-VEGF treatments, and with the known expectations of AV lost without treatment, the data were converted in letters ETDRS chart and here are registered the mean number of letters gained or lost in each group. Ho: Differences between mean measurements before and after are similar H1: Differences between mean measurements before and after are different; Test type: Other — Non-inferiority could be considered if the outcomes were comparable to the most known studies yet published or, in the case of non-treatable disorder, if the acupuncture treatment got to maintain the VA and prevent the losses. There are many known studies with conventional treatment and estimations of the worsening of vision in this pathologies on the time without treatment; p < 0.05, t-test, 1 sided — Using the SPSS program and the non-parametrical technic of Wilcoxon it was determined the p-value. It should be noted that the null hypothesis is that all these eyes should have a zero gain or perhaps a loss in VA at two years of follow-up; From this estimation, it is induced that there are differences in results before and after the treatment; Mean Difference (Final Values) = 15.392 — The datum corresponds to the difference in letters seen between exams at the start and the final examination for all participants. Calculi were made by a Microsoft Excel Descriptive Statistics program; The null hypothesis was no gain or loss in VA. The alternative hypothesis was stabilization or some gain in letters seen over the baseline count.The published studies report a small gain in VA in about a third of participants and only in cases of NV-AMD with conventional treatment, and an expectancy of loss of vision in the other non treated or non-treatable macular diseases. Some of the participants in this trial had had ocular injections without positive change. Non-inferiority in this trial means outcomes of similar magnitude to the known studies

4. Primary Outcome: Number of Eyes That Improved VA From Baseline to End of the Study in Participants With Different Forms of Macular Disease Treated With Acupuncture.
Description: "Improved" was defined as cases that gained in visual acuity (Note: no minimum of letters was defined). "Stable" was defined as visual acuity did not change in the sense of not losing or gaining in the final identification of the optotypes. "Lost" was defined as patients who had a worse vision at the end than at the beginning (e.g., lost visual acuity because the disease continued its course and the treatment was not effective.)
Time Frame: 2 years
Population: Patients with AMD can have both eyes with neovascular AMD or NV-AMD in one of the eyes and No NA-AMD in the fellow.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Groups:
- Acupuncture Group Eyes With NV AMD: Patients with neovascular membrane treated with Acupuncture and massage who improved vision (AV).
  Therapy of Traditional Chinese Medicine (acupuncture and Massage) for 24 months
  Acupuncture has been used for retinal diseases in hospitals of China and in other parts of the world. Some patients in this study had one or both eyes with AMD classified as Neovascular AMD by OCT and retinologist examination. In this group were analyzed 22 eyes of 13 patients, Treatment consists in to put needles on specific points of skin one day each week initially, then with longer spaces of time according to improvement.A total of 11 Chinese needles stainless steel, 25 x 40 were used by manual insertion and left for 12-15 minutes.
  Periocular massage is taught and is practiced daily by the patient him or herself.
Arm/Group | Acupuncture Group Eyes With NV AMD
Number analyzed (Participants) | 13
Number analyzed (eyes) | 22
eyes | 13

5. Secondary Outcome: Percentage of Participants Who Experienced Changes in Vision (Less Opacity, Less Distortion of Lines, Reduction of the Central Shadow)
Description: At study entry, major complaints of patients were collected by survey. Participants also completed a survey at the middle and at the end of the trial. This data is the percentage of participants that reported changes to the main visual complaints that they considered significant in their lives compared with the baseline.
Time Frame: Baseline and end of study (up to 2 years)
Population: All the participants who had a follow up for 24 months filled a survey about their complains and limitation in daily life at the beginning, in the middle time and at the end of the study. The measure is the number of patients who reported improvement.
Measure: Number; unit: percentage of participants improved
Groups:
- Acupuncture Group: Acupuncture and massage Therapy of Traditional Chinese Medicine (acupuncture and Massage) for 24 months
  Acupuncture and massage: Treatment consists in to put needles on specific points of skin one day each week initially, then with longer spaces of time according to improvement. A total of 11 Chinese needles stainless steel, 25 x 40 were used by manual insertion and left for 12-15 minutes.
  Periocular massage is taught and is practiced daily by the patient him or herself.
Arm/Group | Acupuncture Group
Number analyzed (Participants) | 29
percentage of participants improved | 61.45

6. Secondary Outcome: Number of Participants With Adverse Events Both Treatment-related or Not Related to Treatment.
Description: To report this measure the adverse events or risks had to be observed carefully and registered in order to care for the safety and to accomplish regulations of any treatment or medical intervention. For this procedure, the usual risks are some adverse events as moderate to severe pain, bleeding of more than a drop, ecchymosis bigger than 5 millimeters. Deaths and other serious events related or not with the therapeutic procedure, had to be reported.
Time Frame: 2 years
Population: Participants who suffered some adverse event as moderate to severe pain, bleeding of more than a drop, ecchymosis bigger than 5 millimeters. Deaths and other events related or not with the therapeutic procedure.
Measure: Number; unit: participants
Groups:
- Adverse Events: By law, and by the protocol of study the adverse events were monitored. In acupuncture, the risks are not frequent and mainly they can consist of pain in the site of insertion of the needle, minimal bleeding or ecchymosis.
  When the observed adverse events exceed the expectations, should have been reported, i.e., moderate to severe pain, bleeding that is more than a drop, or ecchymosis bigger than 5 millimeters in diameter.
  Similarly, was monitored any trouble related or not with the treatment as serious adverse events and mortality.
Arm/Group | Adverse Events
Number analyzed (Participants) | 29
participants | 0

ADVERSE EVENTS:
Time Frame: Adverse event were carefully observed by 2 years
Description: As adverse event in acupuncture is considered bleeding, haematomas, injury to vital organs
Groups:
- All Study Participants: Intervention: Acupuncture (Traditional Chinese Medicine) and Massage: A total of 11 Chinese needles 25 x 40 were used by manual insertion plus Periocular massage.
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

LIMITATIONS AND CAVEATS:
Participants were limited by lack of knowing and credibility of ophthalmologists in TCM OCTs every 6 months was not possible for some due to the cost. Some patients had independent evaluation and their ophthalmologist appreciated the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No